CLINICAL TRIAL: NCT04858217
Title: Diagnostic Accuracy and Cost-effectiveness Analysis of Serum and Synovial Fluid Markers for the Diagnosis of Periprosthetic Hip and Knee Joint Infections
Brief Title: Periprosthetic Joint Infections: Diagnostic Accuracy and Cost-effectiveness Analysis of Serum and Synovial Markers
Acronym: DECISION
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: 37/2021/Sper/IOR
Record Dates: First submitted 2021-04-08; First posted 2021-04-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Prosthetic Joint Infection
Keywords: prosthetic joint infection; biomarker; synovial fluid; serum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and synovial fluid specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Total joint replacement (TJR) is an increasing effective procedure in orthopedics. However, TJR failure due to aseptic or septic loosening remains an important problem, often due to predisposing factors of the patient, which determine the need to perform a revision surgery. In light of the recent conclusions emerged on the still open problems concerning the diagnostic accuracy of serum and synovial fluid markers in the diagnosis of peri-prosthetic joint infection (PJI), the project aims at evaluating the diagnostic accuracy and cost-effectiveness of the combination of serum and/or synovial markers in the diagnosis of PJI. Through a diagnostic clinical study on patients hospitalized for revision surgery the project would provide evidences on the potentiality of the combination of some markers in accelerating the PJI diagnosis for the best selection of surgical strategy, choosing the suitable cutoff thresholds to mitigate the effect of some factors on markers' discriminatory capability.

DETAILED DESCRIPTION:
Total joint arthroplasties (TJA) are constantly increasing in older and multi-morbid patients; knee and hip joints are the most frequently treated due to high incidence of osteoarthritis in these joints. The indication to TJA is now extended to younger and active patients with high functional demands and longer life expectancy. Because of these, an increase in revision surgeries and a PJI risk is also expected. The type of revision surgery (RS) approach and of antimicrobial treatments is based on the presence or absence of infection: one-stage revision with maintenance/replacement of prosthesis in combination with debridement and irrigation (aseptic RS); and two-stage revision with prosthesis removal, debridement and irrigation, the possible use of a temporary spacer, and the potential reimplantation after weeks or months (septic RS).

Today, PJI remains an important dangerous and devastating complication; it has been reported for hip and knee joints an incidence of 0.2-1.5%, prosthesis failure of 15-25%, revision success rate of 80-95% and annual cost per infection of $20,000-$40,000. The timely and most accurate diagnosis is essential for the correct treatment of PJI as patients undergoing revision need extensive physical, psychological and economic supports. Following the definition and standardization of diagnostic major and minor criteria for PJI by the Musculoskeletal Infection Society (MSIS) an improvement in the diagnosis and treatment of PJI was observed. Recently, the International Consensus Group on PJI revised MSIS criteria defining that patients should be considered to have PJI in the presence of one of the major criteria or three of five minor criteria. Finally, an evidence-based and validated criteria for hip and knee PJI definition to diagnose patients within the preoperative period was published in 2018. Patients with an aggregate score of more than or equal to 6 are considered infected, while a 2-5 score requires the inclusion of intraoperative findings (positive histology, purulence and single positive culture) for confirming or refuting the diagnosis. A 4-5 score is inconclusive, and a score of less than or equal to 3 is not infected.

During the last International Consensus Meeting on Musculoskeletal Infection, various questions on PJI were discussed and among them the working groups (WG) provided recommendations based on limited (4 - due to small numbers) and moderate (12 and 19) levels of evidence: WG4, on which patient-specific factors influence the thresholds for serum and synovial markers in acute and chronic PJI; WG12, on which serum tests have the best diagnostic accuracy for PJI and if the combination of any number of tests increase the diagnostic accuracy; WG19, if the profile of organisms causing surgical site infection or PJI following orthopaedic procedures changed over recent years. The WG4 highlighted that no inflammatory arthritis (IA)-specific factors are known to influence the thresholds for serum and synovial markers in PJIs. It appears that in IA patients there are overlaps in values of synovial markers such as alphadefensin, white blood cell count (sWBC) and C-reactive protein (CRP), limiting their usefulness in differentiating septic from aseptic patients. The WG12 stated that it is evident that diagnosis of PJI cannot be based solely on serological tests and that CRP and erythrocyte sedimentation rate (ESR) are well-researched screening tests and have high sensitivity when used alone. However, the combination of serological tests has shown to improve diagnostic accuracy, but the identification of the optimal combination needs further investigations. Finally, the WG19 recommended to perform further investigations regarding the profile of microorganism with next generation sequencing (NGS), as it may confer significant antibiotic selection implications.

Among pre-operative test on synovial fluid, alpha-defensin showed the highest degree of accuracy in the diagnosis of PJI when measured by laboratory-based immunoassay rather than lateral flow test, suggesting that care must be taken with interpretation of the lateral flow test when relying on its results for the intra-operative diagnosis. Synovial fluid could be tested for other newly markers such calprotectin and cathelicidin LL-37, whose sensitivity and specifity are to be defined or for microbiological tests.

Synovial fluid analysis for WBC and %PMN has high sensitivity and specificity in diagnosing PJI, and it represents an easy and widespread available method. Our meta-analysis evaluated: 1) accuracy in terms of sensitivity and specificity of synovial fluid WBC and %PMN tests in the diagnosis of PJI after total knee (TKA) and hip (THA) arthroplasty; 2) which test yielded superior test performance; and 3) the influence of study characteristics such as anatomic site and threshold value on the diagnostic accuracy of these tests. The meta-analysis results revealed that both synovial fluid WBC and %PMN have a high specificity and sensitivity in detecting PJI, and no clear superiority of one test over the other exists. In addition, an anatomic site effect was demonstrated on sensitivity of synovial fluid %PMN, suggesting that cutoff thresholds should be identified separately for TKA and THA. The differences in bearing surfaces and the possibility of fretting corrosion in dual taper stem designs might substantially alter automated synovial fluid analysis in THA compared to TKA.

The aim of the project is to evaluate the diagnostic accuracy and cost-effectiveness of the combination of serum and/or synovial markers in the pre- or intraoperative (lateral flow test)/post- diagnosis of PJI. To such purpose a clinical diagnostic study on patients hospitalized for revision surgery based on the guidelines of MSIS will be carried out; the combinations of two or more markers with the highest diagnostic accuracies will be identified and evaluated in term of cost-effectiveness towards individual markers whose thresholds are based on the MSIS 2013 ICM. The significance of this research is to provide evidences on the potentiality of the combination of some markers in accelerating the PJI diagnosis for the best selection of surgical strategy to be followed. A prompt diagnosis and recognition of the etiological agent are crucial to define the appropriate antimicrobial therapy and to reduce to a minimum the cases of erroneous diagnosis and of consequent erroneous surgical conduct, with the need for subsequent re-operations, and multiplication of risk for patients and of costs for the health care system.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring hip or knee replacement surgery: i) for 'late' joint prosthesis infection, present for at least 90 days from the date of the arthroplasty (first surgical phase); II) for non-infectious causes (mobilization, wear, instability, misalignment, adverse reactions to local tissues or other aseptic causes), also present for at least 90 days, and which have not had other re-operations on the same joint, and which will be a one-step review;
* Previous clinical data and laboratory and radiological examinations available.

Exclusion Criteria:

* Patients affected by 'early' joint prosthesis infection, with clinical symptom latency of less than 90 days (in this specific subset of patients there is in fact still considerable heterogeneity and little consensus about the diagnostic levels of white blood cell count and percentage of neutrophils).
* Patients suffering from joint prosthesis infection involving joints other than the hip or knee.
* Severe cognitive impairment or psychiatric disorders;
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A maximum number of n = 270 patients who will have to undergo hip or knee prosthetic revision surgery will be enrolled, of which n = 54 for late infection ascertained by previous microbiological analyzes, and n = 216 for prosthetic failure not from infection. Patients will be enrolled in the clinical study only after having signed and dated personally or by the patient's legal representative, the written informed consent. Therefore, enrollment in the study (exclusively of a diagnostic type) will not in any case influence the established diagnostic and therapeutic path.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
White blood cell count (WBC, cells/μL) | 7 days
Erythrocyte sedimentation rate (ESR, mm/hour) | 7 days
C-reactive Protein (CRP, mg/L) | 7 days
D-dimer (ng/ml) | 7 days
IL-6 (pg/ml) | 7 days
Procalcitonin (ng/ml) | 2 months
Soluble Intercellular Adhesion Molecule-1 (sICAM-1, ng/L) | 7 days
Synovial WBC (sWBC, cells/μL) | 7 days
Percentage of polymorphonucleates (%PMM, %) in synovial fluid | 7 days
Synovial C-reactive Protein (sCRP, mg/L) | 7 days
Synovial alpha-defensin (positive or negative) | 7 days
Synovial leukocyte esterase (positive or negative) | 7 days
Synovial IL-6 (pg/ml) | 7 days
Synovial cathelicidin LL-37 (μg/ml) | 7 days
Synovial calprotectin (ng/ml) | 7 days

SECONDARY OUTCOMES:
Serum and synovial biomarkers cut-off for prosthetic joint infections | 2 months
  Test various cut-off values for selected serum and synovial biomarkers for diagnosing PJI.
Assessment of antimicrobial resistances of isolated microrganisms | 2 months
  Bacterial gene sequencing to indentify antimicrobial resistance by Ion AmpliSeqTM Antimicrobial Resistance (AMR) Research Panel.
Assessment of biofilm formation capability of isolated microrganisms | 2 months
  Measure the level of cyclic dimeric bis- (3'-5 ') - guanosine monophosphate (c-di-GMP) which influences biofilm formation by proteomic analysis (MALDI-TOF).

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Giavaresi, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pabinger C, Geissler A. Utilization rates of hip arthroplasty in OECD countries. Osteoarthritis Cartilage. 2014 Jun;22(6):734-41. doi: 10.1016/j.joca.2014.04.009. Epub 2014 Apr 26. PMID 24780823
- [Background] Pabinger C, Lothaller H, Geissler A. Utilization rates of knee-arthroplasty in OECD countries. Osteoarthritis Cartilage. 2015 Oct;23(10):1664-73. doi: 10.1016/j.joca.2015.05.008. Epub 2015 May 29. PMID 26028142
- [Background] Brochin RL, Phan K, Poeran J, Zubizarreta N, Galatz LM, Moucha CS. Trends in Periprosthetic Hip Infection and Associated Costs: A Population-Based Study Assessing the Impact of Hospital Factors Using National Data. J Arthroplasty. 2018 Jul;33(7S):S233-S238. doi: 10.1016/j.arth.2018.02.062. Epub 2018 Feb 22. PMID 29573912
- [Background] Schwarz EM, Parvizi J, Gehrke T, Aiyer A, Battenberg A, Brown SA, Callaghan JJ, Citak M, Egol K, Garrigues GE, Ghert M, Goswami K, Green A, Hammound S, Kates SL, McLaren AC, Mont MA, Namdari S, Obremskey WT, O'Toole R, Raikin S, Restrepo C, Ricciardi B, Saeed K, Sanchez-Sotelo J, Shohat N, Tan T, Thirukumaran CP, Winters B. 2018 International Consensus Meeting on Musculoskeletal Infection: Research Priorities from the General Assembly Questions. J Orthop Res. 2019 May;37(5):997-1006. doi: 10.1002/jor.24293. Epub 2019 Apr 25. PMID 30977537
- [Background] Bonanzinga T, Ferrari MC, Tanzi G, Vandenbulcke F, Zahar A, Marcacci M. The role of alpha defensin in prosthetic joint infection (PJI) diagnosis: a literature review. EFORT Open Rev. 2019 Jan 23;4(1):10-13. doi: 10.1302/2058-5241.4.180029. eCollection 2019 Jan. PMID 30800475
- [Background] Kunutsor SK, Beswick AD, Peters TJ, Gooberman-Hill R, Whitehouse MR, Blom AW, Moore AJ. Health Care Needs and Support for Patients Undergoing Treatment for Prosthetic Joint Infection following Hip or Knee Arthroplasty: A Systematic Review. PLoS One. 2017 Jan 3;12(1):e0169068. doi: 10.1371/journal.pone.0169068. eCollection 2017. PMID 28046049
- [Background] Osmon DR, Berbari EF, Berendt AR, Lew D, Zimmerli W, Steckelberg JM, Rao N, Hanssen A, Wilson WR; Infectious Diseases Society of America. Executive summary: diagnosis and management of prosthetic joint infection: clinical practice guidelines by the Infectious Diseases Society of America. Clin Infect Dis. 2013 Jan;56(1):1-10. doi: 10.1093/cid/cis966. PMID 23230301
- [Background] Parvizi J, Zmistowski B, Berbari EF, Bauer TW, Springer BD, Della Valle CJ, Garvin KL, Mont MA, Wongworawat MD, Zalavras CG. New definition for periprosthetic joint infection: from the Workgroup of the Musculoskeletal Infection Society. Clin Orthop Relat Res. 2011 Nov;469(11):2992-4. doi: 10.1007/s11999-011-2102-9. No abstract available. PMID 21938532
- [Background] Cats-Baril W, Gehrke T, Huff K, Kendoff D, Maltenfort M, Parvizi J. International consensus on periprosthetic joint infection: description of the consensus process. Clin Orthop Relat Res. 2013 Dec;471(12):4065-75. doi: 10.1007/s11999-013-3329-4. Epub 2013 Oct 24. No abstract available. PMID 24155178
- [Background] Parvizi J, Tan TL, Goswami K, Higuera C, Della Valle C, Chen AF, Shohat N. The 2018 Definition of Periprosthetic Hip and Knee Infection: An Evidence-Based and Validated Criteria. J Arthroplasty. 2018 May;33(5):1309-1314.e2. doi: 10.1016/j.arth.2018.02.078. Epub 2018 Feb 26. PMID 29551303
- [Background] Han X, Xie K, Jiang X, Wang L, Wu H, Qu X, Yan M. Synovial fluid alpha-defensin in the diagnosis of periprosthetic joint infection: the lateral flow test is an effective intraoperative detection method. J Orthop Surg Res. 2019 Aug 28;14(1):274. doi: 10.1186/s13018-019-1320-9. PMID 31455372
- [Background] Marson BA, Deshmukh SR, Grindlay DJC, Scammell BE. Alpha-defensin and the Synovasure lateral flow device for the diagnosis of prosthetic joint infection: a systematic review and meta-analysis. Bone Joint J. 2018 Jun 1;100-B(6):703-711. doi: 10.1302/0301-620X.100B6.BJJ-2017-1563.R1. PMID 29855233
- [Background] Suen K, Keeka M, Ailabouni R, Tran P. Synovasure 'quick test' is not as accurate as the laboratory-based alpha-defensin immunoassay: a systematic review and meta-analysis. Bone Joint J. 2018 Jan;100-B(1):66-72. doi: 10.1302/0301-620X.100B1.BJJ-2017-0630.R1. PMID 29305453
- [Background] Wouthuyzen-Bakker M, Ploegmakers JJW, Ottink K, Kampinga GA, Wagenmakers-Huizenga L, Jutte PC, Kobold ACM. Synovial Calprotectin: An Inexpensive Biomarker to Exclude a Chronic Prosthetic Joint Infection. J Arthroplasty. 2018 Apr;33(4):1149-1153. doi: 10.1016/j.arth.2017.11.006. Epub 2017 Nov 13. PMID 29224989
- [Background] Alvand A, Rezapoor M, Parvizi J. The Role of Biomarkers for the Diagnosis of Implant-Related Infections in Orthopaedics and Trauma. Adv Exp Med Biol. 2017;971:69-79. doi: 10.1007/5584_2017_11. PMID 28243953
- [Background] Parvizi J, Gehrke T, Chen AF. Proceedings of the International Consensus on Periprosthetic Joint Infection. Bone Joint J. 2013 Nov;95-B(11):1450-2. doi: 10.1302/0301-620X.95B11.33135. PMID 24151261
- [Background] De Fine M, Giavaresi G, Fini M, Illuminati A, Terrando S, Pignatti G. The role of synovial fluid analysis in the detection of periprosthetic hip and knee infections: a systematic review and meta-analysis. Int Orthop. 2018 May;42(5):983-994. doi: 10.1007/s00264-018-3865-3. Epub 2018 Mar 9. PMID 29523955
- [Background] Hajian-Tilaki K. Sample size estimation in diagnostic test studies of biomedical informatics. J Biomed Inform. 2014 Apr;48:193-204. doi: 10.1016/j.jbi.2014.02.013. Epub 2014 Feb 26. PMID 24582925
- [Background] Moreno et al., Bayesian Cost-Effectiveness Analysis of Medical Treatments. Chapman and Hall/CRC 2019. ISBN 9781138731738